CLINICAL TRIAL: NCT06503003
Title: Non-ablative Diode Laser Therapy for Genitourinary Syndrome of Menopause: A Prospective Study on Efficacy, Safety, and Quality of Life and Sexuality Impact
Acronym: GSMLASER
Status: Recruiting | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Professor, University of Cagliari
Other Study IDs: NP/2022/4057
Record Dates: First submitted 2024-07-05; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: Genitourinary Syndrome of Menopause; Diode laser; Vaginal Atrophy; Menopause; Sexual Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laser Therapy Group: Participants will receive non-ablative dual-wavelength diode laser therapy for Genitourinary Syndrome of Menopause (GSM). The intervention includes three monthly sessions using the Leonardo® Diode laser (Biolitec®) with wavelengths of 980 nm and 1470 nm. Each session lasts about 20 minutes and involves 8 pulses per centimeter along the vaginal canal. Local lidocaine gel is used as an anesthetic. Evaluations occur at baseline, 3 months, and 6 months post-treatment.
  Interventions: Device: Leonardo® Diode laser

INTERVENTIONS:
Device: Leonardo® Diode laser — The intervention involves non-ablative dual-wavelength diode laser therapy for treating Genitourinary Syndrome of Menopause (GSM). This includes three monthly sessions of the Leonardo® Diode laser (Biolitec®), with wavelengths of 980 nm and 1470 nm, delivering 8 pulses per centimeter along the vaginal canal, using local lidocaine gel as an anesthetic. Evaluations are conducted at baseline, 3 months, and 6 months post-treatment.

SUMMARY:
The goal of this observational study is to evaluate the efficacy, safety, and impact on quality of life and sexuality of non-ablative dual-wavelength diode laser treatments in managing Genitourinary Syndrome of Menopause (GSM) in sexually active post-menopausal women who cannot use or have not benefited from local estrogen-based therapies. The main questions it aims to answer are:

Does non-ablative dual-wavelength diode laser therapy improve vaginal dryness, burning sensation, and dyspareunia in post-menopausal women? What is the impact of this therapy on the vaginal health index and sexual function? Researchers will compare the laser-treated group to their baseline measurements to see if non-ablative dual-wavelength diode laser therapy effectively treats GSM.

Participants will:

Undergo three monthly sessions of dual-wavelength diode laser therapy. Participate in follow-up evaluations at three and six months post-treatment. Complete self-assessments of GSM symptoms and questionnaires evaluating sexual function and quality of life at each follow-up.

This study aims to provide preliminary evidence that non-ablative dual-wavelength diode laser therapy is a safe and effective non-hormonal treatment for GSM, addressing a gap in existing treatments for women who cannot use or have not benefited from hormonal therapies.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women aged 45-73 years.
* Sexually active.
* Experiencing physiological amenorrhea for more than 12 months.
* Exhibiting at least one symptom of Genitourinary Syndrome of Menopause (GSM).
* Not using lubricants or hormonal therapy in the previous 6 months.
* Able to provide written informed consent.

Exclusion Criteria:

* Untreated uterine or vulvovaginal cancers.
* Pacemaker or other implanted electrode carriers.
* Severe multi-organ or neurological diseases.
* Active sexually transmitted infections.
* Moderate to severe uterine prolapse.
* Active urinary tract infections.
* Acute or chronic dermatological conditions in the vulvar or vaginal area.
* Active genital herpes.
* Active high-risk Human Papillomavirus (HPV).
* Ischemic tissues, unhealed wounds, sores, or undiagnosed mucosal or epithelial alterations.
* Recent unhealed invasive or ablative surgeries.
* Bleeding disorders or anticoagulant therapy.
* Immunodeficiencies.
* Uncontrolled diabetes.

Ages: 45 Years to 73 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of post-menopausal women aged 45-73 years who are experiencing symptoms of Genitourinary Syndrome of Menopause (GSM). These women are sexually active and have experienced physiological amenorrhea for more than 12 months. The participants have not used lubricants or hormonal therapy in the previous six months. The study targets those who cannot use or have not benefited from local estrogen-based therapies.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Vaginal Dryness | Baseline, 3 months, 6 months after the final laser treatment
  Measurement of the change in vaginal dryness scores using the Visual Analog Scale (VAS). The Visual Analog Scale ranges from 0 to 10, with higher scores indicating worse vaginal dryness.
Change in Burning Sensation | Baseline, 3 months, and 6 months after the final laser treatment
  Measurement of the change in burning sensation scores using the Visual Analog Scale (VAS). The Visual Analog Scale ranges from 0 to 10, with higher scores indicating worse burning sensation.
Change in Pain During Intercourse (Dyspareunia) | Baseline, 3 months, and 6 months after the final laser treatment
  Measurement of the change in pain during intercourse scores using the Visual Analog Scale (VAS). The Visual Analog Scale ranges from 0 to 10, with higher scores indicating worse pain during intercourse.
Change in Vaginal Health Index Score (VHIS) | Baseline, 3 months, and 6 months after the final laser treatment
  Measurement of the change in the Vaginal Health Index Score (VHIS), which examines five aspects of vaginal health: elasticity, fluid volume, pH, epithelial integrity, and moisture. Each component is rated on a scale from 1 (indicating severe vaginal atrophy) to 5 (indicating no clinical signs of vaginal atrophy), with a total score below 15 confirming vaginal atrophy. Higher scores indicate better vaginal health.
Change in Sexual Function | Baseline, 3 months, and 6 months after the final laser treatment
  Measurement of the change in sexual function scores using the Female Sexual Function Index-6 (FSFI-6). The FSFI-6 is a six-item version of the Female Sexual Function Index-19 (FSFI-19) and includes one item from each original domain: desire, arousal, lubrication, orgasm, satisfaction, and pain. Responses range from 0 (no sexual activity) to 5 (optimal function), with higher scores indicating better sexual function. An FSFI-6 score of 19.0 or less indicates sexual dysfunction.
Change in Sexual Quality of Life | Baseline, 3 months, and 6 months after the final laser treatment
  Measurement of the change in scores on the Sexual Quality of Life-Female (SQOL-F) questionnaire. The SQOL-F questionnaire consists of 18 items that assess sexual self-esteem, emotional well-being, and relationship issues. Scores range from 18 to 108, with higher scores indicating better sexual quality of life.
Change in Sexual Function | Baseline, 3 months, and 6 months after the final laser treatment
  Measurement of the change in sexual function scores using the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). The PISQ-12 is a 12-item questionnaire used to evaluate sexual function in patients suffering from urinary incontinence or pelvic organ prolapse. It explores three domains: behavioral-emotive, physical, and partner-related, scored on a 5-point Likert scale from 0 (always) to 4 (never), with reverse scoring for the first four items. Higher scores indicate better sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Angioni, Principal Investigator — University of Cagliari
Locations (1):
- Division of Gynecology and Obstetrics Department of Surgical Sciences, University of Cagliari, Cagliari, Italy, Cagliari, CA, Italy

REFERENCES:
- [Background] Elia D, Gambacciani M, Berreni N, Bohbot JM, Druckmann R, Geoffrion H, Haab F, Heiss N, Rygaloff N, Russo E. Genitourinary syndrome of menopause (GSM) and laser VEL: a review. Horm Mol Biol Clin Investig. 2019 Dec 19;41(1):/j/hmbci.2020.41.issue-1/hmbci-2019-0024/hmbci-2019-0024.xml. doi: 10.1515/hmbci-2019-0024. PMID 31855563
- [Background] Aguiar LB, Politano CA, Costa-Paiva L, Juliato CRT. Efficacy of Fractional CO2 Laser, Promestriene, and Vaginal Lubricant in the Treatment of Urinary Symptoms in Postmenopausal Women: A Randomized Clinical Trial. Lasers Surg Med. 2020 Oct;52(8):713-720. doi: 10.1002/lsm.23220. Epub 2020 Jan 28. PMID 31990089
- [Background] Knight C, Logan V, Fenlon D. A systematic review of laser therapy for vulvovaginal atrophy/genitourinary syndrome of menopause in breast cancer survivors. Ecancermedicalscience. 2019 Dec 12;13:988. doi: 10.3332/ecancer.2019.988. eCollection 2019. PMID 32010212
- [Background] Samuels JB, Garcia MA. Treatment to External Labia and Vaginal Canal With CO2 Laser for Symptoms of Vulvovaginal Atrophy in Postmenopausal Women. Aesthet Surg J. 2019 Jan 1;39(1):83-93. doi: 10.1093/asj/sjy087. PMID 29726916
- [Background] Karcher C, Sadick N. Vaginal rejuvenation using energy-based devices. Int J Womens Dermatol. 2016 Jun 21;2(3):85-88. doi: 10.1016/j.ijwd.2016.05.003. eCollection 2016 Sep. PMID 28492016
- [Background] Eder SE. Early effect of fractional CO2 laser treatment in Post-menopausal women with vaginal atrophy. Laser Ther. 2018 Mar 31;27(1):41-47. doi: 10.5978/islsm.18-OR-04. PMID 29795970
- [Background] Gambacciani M, Levancini M, Russo E, Vacca L, Simoncini T, Cervigni M. Long-term effects of vaginal erbium laser in the treatment of genitourinary syndrome of menopause. Climacteric. 2018 Apr;21(2):148-152. doi: 10.1080/13697137.2018.1436538. Epub 2018 Feb 13. PMID 29436235
- [Background] Angioni S, Mais V, Pontis A, Peiretti M, Nappi L. First case of prophylactic salpingectomy with single port access laparoscopy and a new diode laser in a woman with BRCA mutation. Gynecol Oncol Case Rep. 2014 May 19;9:21-3. doi: 10.1016/j.gynor.2014.05.002. eCollection 2014 Aug. PMID 25426409
- [Background] Angioni S, Pontis A, Sorrentino F, Nappi L. Bilateral salpingo-oophorectomy and adhesiolysis with single port access laparoscopy and use of diode laser in a BRCA carrier. Eur J Gynaecol Oncol. 2015;36(4):479-81. PMID 26390708
- [Background] Nappi L, Angioni S, Sorrentino F, Cinnella G, Lombardi M, Greco P. Anti-Mullerian hormone trend evaluation after laparoscopic surgery of monolateral endometrioma using a new dual wavelengths laser system (DWLS) for hemostasis. Gynecol Endocrinol. 2016;32(1):34-7. doi: 10.3109/09513590.2015.1068754. Epub 2015 Aug 28. PMID 26359914
- [Background] Nappi L, Pontis A, Sorrentino F, Greco P, Angioni S. Hysteroscopic metroplasty for the septate uterus with diode laser: a pilot study. Eur J Obstet Gynecol Reprod Biol. 2016 Nov;206:32-35. doi: 10.1016/j.ejogrb.2016.08.035. Epub 2016 Aug 31. PMID 27632410
- [Background] Nappi L, Sorrentino F, Angioni S, Pontis A, Litta P, Greco P. Feasibility of hysteroscopic endometrial polypectomy using a new dual wavelengths laser system (DWLS): preliminary results of a pilot study. Arch Gynecol Obstet. 2017 Jan;295(1):3-7. doi: 10.1007/s00404-016-4232-5. Epub 2016 Nov 11. PMID 27834002
- [Background] Esteban Manchado B, Lopez-Yarto M, Fernandez-Parra J, Rodriguez-Oliver A, Gonzalez-Paredes A, Lagana AS, Garzon S, Haimovich S. Office hysteroscopic metroplasty with diode laser for septate uterus: a multicenter cohort study. Minim Invasive Ther Allied Technol. 2022 Mar;31(3):441-447. doi: 10.1080/13645706.2020.1837181. Epub 2020 Oct 22. PMID 33090039
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Maasoumi R, Lamyian M, Montazeri A, Azin SA, Aguilar-Vafaie ME, Hajizadeh E. The sexual quality of life-female (SQOL-F) questionnaire: translation and psychometric properties of the Iranian version. Reprod Health. 2013 May 5;10:25. doi: 10.1186/1742-4755-10-25. PMID 23642126
- [Background] Fahndrich E, Linden M. [Reliability and validity of the Visual Analogue Scale (VAS) (author's transl)]. Pharmacopsychiatria. 1982 May;15(3):90-4. doi: 10.1055/s-2007-1019515. German. PMID 7100262
- [Background] Bachmann GA, Phillips NA. Vaginal health prescription: possible next step in the management of genitourinary syndrome of menopause. Menopause. 2015 Feb;22(2):127-8. doi: 10.1097/GME.0000000000000414. No abstract available. PMID 25549067
- [Background] Dargie E, Holden RR, Pukall CF. The Vulvar Pain Assessment Questionnaire: Factor Structure, Preliminary Norms, Internal Consistency, and Test-Retest Reliability. J Sex Med. 2017 Dec;14(12):1585-1596. doi: 10.1016/j.jsxm.2017.10.072. PMID 29198513
- [Derived] Vitale SG, Saponara S, Succu AG, Sicilia G, Martsidis K, D'Alterio MN, Angioni S. Efficacy and Safety of Non-Ablative Dual Wavelength Diode Laser Therapy for Genitourinary Syndrome of Menopause: A Single-Center Prospective Study. Adv Ther. 2024 Dec;41(12):4617-4627. doi: 10.1007/s12325-024-03004-7. Epub 2024 Oct 29. PMID 39470875